CLINICAL TRIAL: NCT05873634
Title: HeartShare Deep Phenotyping Study
Brief Title: HeartShare: Combining Omics, Deep Phenotyping, and Electronic Health Records for Heart Failure Subtypes and Treatment Targets
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Mayo Clinic (Other); University of California, Davis (Other); Wake Forest University Health Sciences (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sanjiv Shah, Stone Endowed Professor of Medicine, Director of Research, Bluhm Cardiovascular Institute, Principal Investigator, HeartShare Data Translation Center, Northwestern University
Other Study IDs: STU00217900; U54HL160273 (NIH)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Plasma, serum, RNA, DNA, urine, saliva, and stool samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFpEF: Participants with HFpEF
- Non-HFpEF: Participants without HFpEF

SUMMARY:
HeartShare is a comprehensive study of heart failure, a common and serious medical condition which occurs when the heart is unable to keep up with the demands of the body, resulting in shortness of breath, fluid retention, and fatigue. HeartShare aims to better classify heart failure into subtypes to help develop more personalized treatments for patients, with the hope that this will improve the lives of heart failure patients. To do this, HeartShare is bringing together a large amount of data (including images, such as heart ultrasounds and MRIs and molecular data from the blood, such as genetics) from previously conducted studies and electronic health records, and is gathering new data through participants enrolled in the HeartShare Deep Phenotyping Study.

ELIGIBILITY:
Inclusion Criteria:

HF Inclusion Criteria (HeartShare Registry)

1. Age ≥30 years.
2. Prior diagnosis of HF in the EHR (any left ventricular ejection fraction).

Non-HF Group Inclusion Criteria (HeartShare Registry)

1. Age ≥30 years.
2. No known prior diagnosis of HF or use of loop diuretics.
3. No known prior history of BNP >100 pg/ml or NTproBNP >300 pg/ml, if prior laboratory tests are available in the EHR.

HFpEF Inclusion Criteria (HeartShare Deep Phenotyping Cohort)

1. Age ≥30 years.
2. Left ventricular ejection fraction ≥50% measured by echocardiography.
3. Definition of HFpEF: signs and symptoms of HF, NYHA functional class II-IV, and at least one of the following:

   1. Elevated BNP (≥75 pg/ml in sinus rhythm or ≥225 pg/ml in atrial fibrillation/flutter) or NTproBNP (≥225 pg/ml in sinus rhythm or ≥675 in atrial fibrillation/flutter) at baseline. Choice of BNP or NTproBNP is based on availability at each clinical center.
   2. Prior HF hospitalization (primary reason for the hospitalization is HF with elevated natriuretic peptide levels [using the thresholds listed above], requiring IV diuresis for HF, or pulmonary edema or pulmonary vascular congestion on chest radiography).
   3. Elevated pulmonary capillary wedge pressure (PCWP) at rest (≥15 mmHg) or during exercise (≥25 mmHg for supine exercise or PCWP/cardiac output ratio ≥2 mmHg/L/min for upright exercise).
   4. Elevated H2FPEF score26 (≥5) or HFA-PEFF27 score (≥5).

Non-HFpEF Group Inclusion Criteria (HeartShare Deep Phenotyping Cohort)

1. Age ≥30 years.
2. Left ventricular ejection fraction ≥50% measured by echocardiography.
3. No known prior diagnosis of HF or use of diuretics for fluid management.
4. No known prior history of BNP ≥75 pg/ml or NTproBNP ≥225 pg/ml, if prior laboratory tests are available in the EHR.
5. BNP <75 pg/ml or NTproBNP <225 pg/ml at the time of screening. Choice of BNP or NTproBNP is based on availability at each clinical center.

Exclusion Criteria:

Exclusion Criteria (HeartShare Registry) The following exclusion criteria apply to both HF and non-HF group participants, unless otherwise indicated.

1. For non-HF group: any prior known left ventricular ejection fraction <50%.
2. Prior history of solid organ transplantation.
3. Prior history of mechanical circulatory support.
4. Prior history of non-cardiac cirrhosis.
5. Inability to provide written consent to the study.

Exclusion Criteria (HeartShare Deep Phenotyping Cohort) The following exclusion criteria apply to both HFpEF and non-HFpEF group participants, unless otherwise indicated.

1. Life expectancy estimated to be < 1 year.
2. Primary cardiomyopathy (including amyloid, hypertrophic cardiomyopathy, cardiac sarcoidosis, hemochromatosis, or other infiltrative cardiomyopathies) or pulmonary arterial hypertension (WHO Group I, III, or IV pulmonary hypertension).
3. Any prior known left ventricular ejection fraction <40%, except if this occurred only in the setting of an acute tachycardia episode (e.g., acute atrial fibrillation).
4. Clinically significant valvular heart disease defined as:

   1. Moderate to greater aortic stenosis, pulmonic stenosis, or tricuspid stenosis.
   2. Any mitral stenosis.
   3. Moderate or greater aortic regurgitation.
   4. Greater than moderate mitral regurgitation.
5. Any planned cardiac surgery or cardiac intervention in the next 3 months.
6. Alternative primary reason for symptoms of shortness of breath and exercise intolerance in HFpEF participants in the opinion of the enrolling investigator.
7. Cardiac surgery, acute coronary syndrome, percutaneous coronary intervention, stroke, transient ischemic attack, or carotid intervention in the preceding 6 months prior to enrollment.
8. Known symptomatic epicardial coronary artery disease that is not revascularized.
9. Any non-elective hospitalization in the preceding 2 weeks.
10. Prior history of solid organ transplantation.
11. Prior history of chronic infection (HIV, hepatitis C, hepatitis B, tuberculosis) unless treated and not clinically active in the opinion of the enrolling investigator.
12. Prior history of mechanical circulatory support.
13. Prior history of non-cardiac cirrhosis.
14. Estimated GFR <20 ml/min/1.73m2 or currently on dialysis.
15. Any condition that may preclude participation or adherence to the study protocol, in the opinion of the enrolling investigator.
16. Inability to provide written consent to the study.
17. Current acute decompensated heart failure.
18. Currently pregnant.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 30 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Heart Failure with Preserved Ejection Fraction (HFpEF) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern University; Svati Shah, MD, MHS, Study Chair — Duke University; Javed Butler, MPH, MBA, Study Chair — Baylor Scott and White Health
Locations (6):
- United States (6):
  - University of California Davis, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - Mass General Brigham, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania